CLINICAL TRIAL: NCT06930833
Title: FRAILTY Classification Algorithm for the Corsano CARDIOWATCH 287-2: a Development and Validation Study
Acronym: FRAILTY-CW2
Status: Not yet recruiting | Type: Observational
Sponsor: Corsano Health B.V. (Industry)
Responsible Party: Sponsor
Other Study IDs: FRAILTY
Record Dates: First submitted 2025-04-09; First posted 2025-04-16 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Cardiac Arrythmias; Valve Heart Disease; Cardiac Ischemia
Keywords: Frailty; 6-minute walking test; G8-score; wristband; wearable; remote monitoring; cardiac surgical interventions
MeSH Terms: conditions — Heart Valve Diseases; Coronary Artery Disease; Frailty

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing cardiac surgical intervention: Patients ≥ 70 years of age who are scheduled to undergo aortic valve replacement, mitral valve repair with MitraClip, implantation of a pacemaker or percutaneous coronary intervention (PCI) at the Reinier de Graaf Gasthuis Cardiology department.
  Interventions: Device: Corsano CardioWatch 287-2

INTERVENTIONS:
Device: Corsano CardioWatch 287-2 — Eligible patients are asked to wear the Corsano CardioWatch 287-2 for 6 days, of which 3 days approximately 2 weeks before the procedure and 3 days approximately 2 months after the procedure.

SUMMARY:
The FRAILTY-CARDIOWATCH study is investigating how well the Corsano CardioWatch 287-2, a wrist-worn medical device, can classify frailty in patients. Frailty is a condition often seen in older adults, characterized by decreased strength, endurance, and overall health, which can make individuals more vulnerable to illness or injury. The goal of this study is to develop an algorithm that can accurately assess frailty using the device. In phase 1 of the study, data will be collected from patients aged 70 or older who are scheduled for heart-related procedures, such as valve replacements or pacemaker implantation.

The study aims to compare the frailty classifications of the CardioWatch with two established methods: the Geriatric 8 (G8) questionnaire and the FRAIL scale. It will also compare the CardioWatch with the 6-minute walk test. Patients will wear the CardioWatch for six days-three days before their procedure and three days after-and complete the G8, FRAIL, and 6-minute walk tests. The collected data will help develop and train the frailty classification algorithm.

The main focus is to evaluate how well the frailty classifications from the CardioWatch match those from the other tests. This research could potentially lead to a more accurate and continuous way to monitor frailty in patients using wearable technology.

DETAILED DESCRIPTION:
Rationale:

Wrist wearables have the potential to continuously and accurately classify frailty. The Corsano CardioWatch 287-2 is such a medical device with that potential. The collection of clinical data is required to develop, train and validate an algorithm to classify frailty for the Corsano CardioWatch 287-2. The FRAILTY-CARDIOWATCH study consists of two phases, of which only phase 1 (data collection and algorithm development and training) will be addressed in this protocol.

Primary Objective:

The main objective is to determine the agreement of the frailty classification between the Corsano CardioWatch and the gold standard Geriatric 8 (G8) questionnaire as well as the FRAIL scale.

Secondary objectives:

The secondary objective is to determine the agreement of the frailty classification between the Corsano CardioWatch and the 6-minute walk test (6MWT).

Study population:

Patients ≥ 70 years of age who are scheduled to undergo aortic valve replacement, mitral valve repair with MitraClip, implantation of a pacemaker or percutaneous coronary intervention (PCI) at the Reinier de Graaf Gasthuis Cardiology department.

Study design:

Patients are asked to undergo a G8 assessment, FRAIL scale assessment, 6MWT and wear the Corsano CardioWatch 287-2 for 6 days; of which 3 days approximately 2 weeks before the procedure, and 3 days approximately 2 months after the procedure. Collected data of 20 patients will be used to develop and train a frailty classification algorithm for the Corsano CardioWatch 287-2 (phase I).

Main study parameters/endpoints:

Accuracy of the frailty classifications between the G8 assessment or FRAIL scale and the frailty algorithm of Corsano CardioWatch 287-2.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 70 years old
* Be able to provide consent
* Be scheduled to undergo one of the following procedures:

  * Aortic valve replacement
  * Mitral valve repair with MitraClip
  * Implantation of a pacemaker
  * Percutaneous coronary intervention (PCI)

Exclusion Criteria:

* Unable to wear the Corsano CardioWatch 287-2 due to reasons such as allergic reactions, wounds, amputations etc.;
* Unable or unwilling to sign informed consent;
* Significant mental or cognitive impairment;
* Cardiovascular disease where heart rate is not measurable (e.g. LVAD)

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients ≥ 70 years of age who are scheduled to undergo aortic valve replacement, mitral valve repair with MitraClip, implantation of a pacemaker or percutaneous coronary intervention (PCI) at the Reinier de Graaf Gasthuis Cardiology department.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Frailty score agreement between Geriatric-8 questionnaire and CardioWatch 287-2 | From start to end of first CardioWatch 287-2 measurement (~2 week prior to surgery) and from start to end of second CardioWatch 287-2 measurement ('~2 months after surgery)
  G8 questionnaire: when a G8 score ≤ 14 is obtained the patient is considered as frail. When a G8 score > 14 is obtained the patient is considered as non-frail
  The following parameters will be calculated:
  * Accuracy: the proportion of correctly classified frailty stages compared to the total number of frailty stages. This accuracy will be calculated for every participant separately and will thereafter be averaged over all patients.
    o Accuracy: (TP + TN) / (TP + TN + FP + FN)
  * For comparing the G8 score outcomes and the CardioWatch frailty scores the (frail vs. non-frail) the following parameters will be calculated:
    * Specificity: TN / (TN + FP)
    * Sensitivity: TP / (TP + FN)
Frailty score agreement between FRAIL questionnaire and CardioWatch 287-2 | From start to end of first CardioWatch 287-2 measurement (~2 week prior to surgery) and from start to end of second CardioWatch 287-2 measurement ('~2 months after surgery)
  FRAIL score: when a FRAIL score ≥ 3 is obtained the patient is considered as frail.
  When a FRAIL score of 1-2 is obtained the patient is considered as pre-frail, and when a FRAIL score of 0 is obtained the patient is considered as non-frail.
  The following parameters will be calculated:
  * Accuracy: the proportion of correctly classified frailty stages compared to the total number of frailty stages. This accuracy will be calculated for every participant separately and will thereafter be averaged over all patients.
    o Accuracy: (TP + TN) / (TP + TN + FP + FN)
  * For comparing the FRAIL score outcomes and the CardioWatch frailty scores (frail, pre-frail and non-frail) the following parameters will be calculated for every outcome possibility (CardioWatch: frail; pre-frail; non-frail) and participant separately and will thereafter be averaged per outcome possibility over all patients:
    * Specificity: TN / (TN + FP)
    * Sensitivity: TP / (TP + FN)

SECONDARY OUTCOMES:
Frailty score agreement between 6-minute walking test and CardioWatch 287-2 | From start to end of first CardioWatch 287-2 measurement (~2 week prior to surgery) and from start to end of second CardioWatch 287-2 measurement ('~2 months after surgery)
  Participants will be categorized based on the 6MWT. If the 6MWT is less than 300 meters, the participant is categorized as low endurance (LE). If the 6MWT is greater than 300 meters, the participant is classified as normal endurance (NE). The 300 meter cut off point ismchosen because it is widely used in literature.
  The following parameters will be calculated for every participant separately and will thereafter be averaged over all patients:.
  * Accuracy: (TP + TN) / (TP + TN + FP + FN)
  * Specificity: TN / (TN + FP)
  * Sensitivity: TP / (TP + FN)

CONTACTS AND LOCATIONS:
Overall Officials: Mariska van Vliet, MD, PhD, Principal Investigator — Reinier de Graaf Groep
Locations (1):
- Reinier de Graaf Gasthuis, Delft, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No